CLINICAL TRIAL: NCT03597711
Title: Comparison of 24G Versus 26G Peripheral Intravenous Safety Cannula and a 24G Non Safety Cannula in a Population of Neonates <32 Weeks Gestation and <1.5Kg Birthweight
Brief Title: Comparing the Effectiveness of a Safety Intravenous Cannula With a Standard Intravenous Cannula in Neonates
Acronym: LittleReed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R04615
Record Dates: First submitted 2018-06-14; First posted 2018-07-24 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Preterm Infant
Keywords: Peripheral Intravenous cannulation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Once consent is obtained, patients will be randomized to either 24G non-safety cannula, 24G safety or 26G safety cannula. Each patient can enter the study a maximum of three times providing 90 episodes of cannulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IVCannulation 24G non-safety cannula (Active Comparator): Peripheral Intravenous cannulation using 24G non-safety cannula
  Interventions: Device: IVcannulation
- IVCannulation 26G safety cannula (Active Comparator): Peripheral Intravenous cannulation using 26G safety cannula
  Interventions: Device: IVcannulation
- IVCannulation 24G safety cannula (Active Comparator): Peripheral Intravenous cannulation using 24G safety cannula
  Interventions: Device: IVcannulation

INTERVENTIONS:
Device: IVcannulation — Peripheral venous cannulation is a common procedure on neonatal NICU, especially in preterm infants
  Other Names: 24G non-safety cannula,26G safety cannula,24G safety cannula

SUMMARY:
A smaller caliber of intravenous cannulae decreases the number of thrombi and phlebitis and improves the duration of peripheral access. It also reduces the incidence of extravasation. 26G cannulae are easier to insert and reduce the number of attempts for cannulation. Safety cannulae are equivalent in terms of durability and ease of insertion, additionally providing a reduction in needle stick injury amongst healthcare professionals and patients.

The goal of this study is to reduce the number of peripheral line insertions and resulting complications in neonates.

The Investigators propose to compare 24G safety and 26G safety cannulae with non-safety 24G cannulae in infants < 32 weeks Gestation and < 1.5 kg weight in terms of length of stay of cannula, ease of insertion and rates of complications such as thrombosis, phlebitis and extravasation.

The Investigators will also evaluate the frequency of needle stick injury to staff and patients in the course of the study.

DETAILED DESCRIPTION:
Peripheral venous cannulation is a common procedure on neonatal NICU. Insertion of peripheral cannulae in neonates is a painful and stressful procedure (5) and it is therefore desirable to minimize the number of procedures by increasing the survival time of each cannula. The incidence of phlebitis is variously described as 20 - 80% (2). Failure of venous access is often due to thrombi, phlebitis and extravasation. Mechanical phlebitis can be avoided by using the smallest gauge cannula capable of delivering the prescribed drug. (1) Mechanical phlebitis occurs where there is movement of a foreign object (cannula) within a vein causing friction and subsequent inflammation(3). Success rates for cannulation depend on a range of factors including the clinician's experience, gauge of cannula and infants weight as well as the condition of veins. Median survival of 24G Teflon intravenous cannulae was described as 40 hours in one study (4). There are few studies on the appropriate sizing of intravenous cannulae in children.

Flow rates for intravenous devise vary greatly depending on the manufacturer. Flow rates for 24G cannulae are 13 - 29 ml/min. The 26G cannulae achieve flow rates of 13 -19 ml/min which is adequate for use on NICU. The most commonly used devise on NICU SMH are 24G cannulae with a flow rates between13ml/min and 25 ml/min depending on manufacturer.

In this study the proposed non-safety 24 G cannula achieves a flow rate of 25 ml/min whereas the safety 24G and 26 G cannula achieve 22ml/ min and 15ml/min respectively.

Within the EU safety devices are mandatory since 2010 (6). Needle stick injuries during venepuncture pose a risk for healthcare professionals and other staff due to the transmission of blood borne pathogens such as Hepatitis B, Hepatitis C and HIV. This has cost implications for the NHS.

Safety cannulae in both 24 and 26 G have been trialed on the investigator's NICU in 2017 and are felt to be an important addition providing both safe and reliable cannulation. The design of the safety cannula is very similar to cannulae already used on the unit and handling does not require change in practice.

Due to the winged design of both safety and non-safety cannulae fixation of the line post insertion can be standardized.

ELIGIBILITY:
Inclusion Criteria:

* Neonates < 32 Gestation
* < 1.5 kg weight
* Admitted to NICU,St Mary's Hospital Manchester.

Exclusion Criteria:

.Neonates with severe skin conditions such as Epidermolysis Bullosa.

* Infants of > 32 weeks Gestation
* > 1.5 kg in birth weight. .Known difficult venous access (clinical decision). .Expected transfer to different neonatal or paediatric unit within 24hr of intended cannulation.

.Patients considered for reorientation of care or palliative care. .Infants previously recruited to the study who had a total of 3 episodes of randomization.

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
length of stay of cannula | Maximum of a week
  How long the cannula continues to work

SECONDARY OUTCOMES:
ease of insertion | Maximum of a week
  How easy or difficult staff find the cannula to insert
rates of complications | Average of a week
  thrombosis, phlebitis and extravasation

OTHER OUTCOMES:
frequency of needle stick injury | At time of Insertion
  To staff and patients

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawleletz, Principal Investigator — Manchester University Foundation Trust, Manchester
Locations (1):
- Neonatal Intensive Care Unit, St Mary's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panadero A, Iohom G, Taj J, Mackay N, Shorten G. A dedicated intravenous cannula for postoperative use effect on incidence and severity of phlebitis. Anaesthesia. 2002 Sep;57(9):921-5. doi: 10.1046/j.1365-2044.2002.02786.x. PMID 12190760
- [Background] Stokowski G, Steele D, Wilson D. The use of ultrasound to improve practice and reduce complication rates in peripherally inserted central catheter insertions: final report of investigation. J Infus Nurs. 2009 May-Jun;32(3):145-55. doi: 10.1097/NAN.0b013e3181a1a98f. PMID 19444022
- [Background] Gupta P, Rai R, Basu S, Faridi MM. Life span of peripheral intravenous cannula in a neonatal intensive care unit of a developing country. J Pediatr Nurs. 2003 Aug;18(4):287-92. doi: 10.1016/s0882-5963(03)00052-6. PMID 12923741